CLINICAL TRIAL: NCT02799290
Title: The Effect of Adipose Tissue Extract and Platelet-rich Plasma on Split-thickness Donor Site Wound Healing. A Comparative Study
Brief Title: Adipose Tissue Extract and Platelet-rich Plasma Use for Wound Healing
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tampere University (Other)
Responsible Party: Principal Investigator, Jenny Lopez, Medical Doctor, Tampere University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R15034
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Results first posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2020-12

CONDITIONS: Wound Healing Disturbance of

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CONTROL (No Intervention): No intervention
- ADIPOSE TISSUE EXTRACT (Experimental): Adipose Tissue extract application
  Interventions: Biological: ADIPOSE TISSUE EXTRACT
- PLATELET-RICH PLASMA GEL (Experimental): PLATELET RICH PLASMA GEL APPLICATION
  Interventions: Biological: PLATELET-RICH PLASMA GEL

INTERVENTIONS:
Biological: ADIPOSE TISSUE EXTRACT — Adipose tissue extract is obtained on site with lipoaspirate adipose tissue prepared though incubation and filtration
  Other Names: ATE
  Arms: ADIPOSE TISSUE EXTRACT
Biological: PLATELET-RICH PLASMA GEL — Autologous platelet rich plasma is obtained onsite and activated following commercial kit instructions
  Other Names: PRP
  Arms: PLATELET-RICH PLASMA GEL

SUMMARY:
Adipose Tissue Extract (ATE) has been found to be an autologous source of growth factors with proven in vitro angiogenic and adipogenic properties.It is obtained by a simple lipoaspirate procedure. We sought to compare the effect of ATE with another known source, platelet-rich plasma to compare the wound healing characteristics on skin graft donor sites.

DETAILED DESCRIPTION:
The investigators enrolled 24 participants with an indication for skin graft. Two or more split-thickness grafts are harvested per patient, one serving as control and the other as experimental. The experimental sites were covered with either autologous PRP gel or ATE prepared in the OR, which was selected in an unblinded manner due to surgical theater convenience. However, donor sites were randomized through a computer generator. Covered with a semiocclusive film, wounds were separated and followed up on days 3,5,7,10,14 for wound healing and 30 and 60 for scar evaluation. Digital photography and specto-photocutometry was employed to know the hemoglobin and melanin content of the wounds, and custom-made software was used to calculate the percentage of wound re-epithelialization.

ELIGIBILITY:
Inclusion Criteria:

* donor site indication

Exclusion Criteria:

* immunosupressive states
* terminal renal insufficiency
* pregnancy
* coagulation dyscrasias
* active infection in donor site

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timo Ylikomi, PhD, Study Director — Tampere University
Locations (1):
- Jenny Lopez, Ilkka Kaartinen, Tampere, Pirkanmaa, Finland

IPD SHARING:
Plan to Share IPD: No
If required, individual data can be shown

REFERENCES:
- [Result] Sarkanen JR, Kaila V, Mannerstrom B, Raty S, Kuokkanen H, Miettinen S, Ylikomi T. Human adipose tissue extract induces angiogenesis and adipogenesis in vitro. Tissue Eng Part A. 2012 Jan;18(1-2):17-25. doi: 10.1089/ten.TEA.2010.0712. Epub 2011 Oct 4. PMID 21902602
- [Result] Sarkanen JR, Ruusuvuori P, Kuokkanen H, Paavonen T, Ylikomi T. Bioactive acellular implant induces angiogenesis and adipogenesis and sustained soft tissue restoration in vivo. Tissue Eng Part A. 2012 Dec;18(23-24):2568-80. doi: 10.1089/ten.TEA.2011.0724. Epub 2012 Aug 17. PMID 22738319

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: donor site
Groups:
- CONTROL: No treatment
Period: Overall Study
Arm/Group | CONTROL | ADIPOSE TISSUE EXTRACT | PLATELET-RICH PLASMA GEL
Started | 24; 28 donor site | 13; 15 donor site | 11; 13 donor site
Completed | 24; 28 donor site | 13; 15 donor site | 11; 13 donor site
Not Completed | 0; 0 donor site | 0; 0 donor site | 0; 0 donor site

BASELINE CHARACTERISTICS:
Population: Wound healing characteristics of donor sites in time
Groups:
- Total: Total of all reporting groups
Arm/Group | CONTROL | ADIPOSE TISSUE EXTRACT | PLATELET-RICH PLASMA GEL | Total
Number analyzed (Participants) | 24 | 13 | 11 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 10 | 2 | 25
  >=65 years | 11 | 3 | 9 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (16.82) | 56.07 (16.57) | 62.45 (17.23) | 59 (16.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 3 | 12
  Male | 18 | 10 | 8 | 36

OUTCOME MEASURES:

1. Primary Outcome: Wound Re-epithelization
Description: observational-digital photography with specialized custom-made software
Time Frame: 30 days
Population: Measured as a whole per group as mean and standard deviation of group and not participant healing.
Measure: Number; unit: days
Arm/Group | CONTROL | ADIPOSE TISSUE EXTRACT | PLATELET-RICH PLASMA GEL
Number analyzed (Participants) | 24 | 13 | 11
days | 12.34 | 10.27 | 11.33

2. Secondary Outcome: Scar Properties
Description: Vancouver Manchester modified scar scale Minimum value 0 maximum value 14 Higher scores mean worse outcome (Scale analyzes 5 wound characteristics in a numeric scale, where 0 is the best scar outcome and 14 the worst. These characteristics are wound: pigmentation, height, vascularity, contour, texture and brightness.) See scale below Vascularity Normal 0 Pink 1 Red 2 Purple 3 Pigmentation Normal 0 Hypopigmentation 1 Hyperpigmentation 2
  Height Flat 0 Depressed1 Elevated 2 Matte vs. shine Shine 0 Matte 1 Contour Forms part of the adjacent skin 0 Small indentation or invagination 1 Hypertrophic 2 Keloid 3 Texture Normal 0 Barely palpable 1 Rough 2 Indented 3
Time Frame: 30 and 60 days
Population: Modified Vancouver/Manchester scar scale at 30 days
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- CONTROL ATE; CONTROL PRP: No treatment
Arm/Group | CONTROL ATE | ADIPOSE TISSUE EXTRACT | PLATELET-RICH PLASMA GEL | CONTROL PRP
Number analyzed (Participants) | 13 | 13 | 11 | 11
units on a scale
  DAY 30 | 8.13 (2.795) | 4.86 (2.13) | 6.46 (2.53) | 6.85 (2.23)
  DAY 60 | 5.66 (2.8) | 2.4 (2.2) | 3.23 (2.4) | 5.69 (2.2)

3. Secondary Outcome: Oxygenated Hemoglobin
Description: Spectophotocutometry measurements with specialized digital camera and software analysis measured in estimated concentration changes (ECC). ECC is a ratio of light reflected hemoglobin chromofore on a special diode light camera. The ratio is between the scar and the adjacent normal skin and is an arbitrary scale previously published. From 0 to 1, where 1 are values closest to the adjacent healthy unscarred skin.
Time Frame: day 30 and 60
Measure: Mean (Standard Deviation); unit: Arbitrary units
Arm/Group | CONTROL | ADIPOSE TISSUE EXTRACT | PLATELET-RICH PLASMA GEL | CONTROL PRP
Number analyzed (Participants) | 13 | 13 | 11 | 11
Arbitrary units
  Day 30 | 0.36 (0.18) | 0.20 (0.22) | 0.24 (0.31) | 0.28 (0.25)
  Day 60 | 0.18 (0.30) | 0.19 (0.11) | 0.09 (0.17) | 0.01 (0.16)

4. Secondary Outcome: Melanin Concentration in Wound
Description: Melanin concentration measured by spectophotocutometry and analyzed by computer software and represented in estimated concentration changes (ECC), as explained above is an arbitrary ratio between the light absorbance between the scar and the adjacent healthy (unscarred skin) for the melanin chromofore.
Time Frame: day 30 and 60
Measure: Mean (Standard Deviation); unit: Arbitrary units
Groups:
- PRP Control: no treatment
Arm/Group | CONTROL | ADIPOSE TISSUE EXTRACT | PLATELET-RICH PLASMA GEL | PRP Control
Number analyzed (Participants) | 13 | 13 | 11 | 11
Arbitrary units
  DAY 30 | 0.02 (0.02) | 0.03 (0.03) | 0.03 (0.03) | 0.03 (0.03)
  DAY 60 | 0.01 (0.01) | 0.02 (0.04) | 0.02 (0.02) | 0.03 (0.03)

ADVERSE EVENTS:
Time Frame: 60 days
Arm/Group | CONTROL | ADIPOSE TISSUE EXTRACT | PLATELET-RICH PLASMA GEL
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/13 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/13 | 0/11
Other Adverse Events (participants affected / at risk) | 0/24 | 0/13 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes